CLINICAL TRIAL: NCT05030740
Title: Thoracic Aortic Stent-graft Study for the Treatment of Thoracic Aortic Pathologies - Assessment of the Relay Plus and Relay NBS Plus Stent-graft
Brief Title: French Assessment of the Relay Plus and Relay NBS Plus Thoracic Stent-Graft
Status: Completed | Type: Observational
Sponsor: Vascutek Ltd. (Industry)
Collaborators: Federation of Medical Specialties (Other)
Responsible Party: Sponsor
Other Study IDs: EFER
Record Dates: First submitted 2021-08-18; First posted 2021-09-01 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Pathology of the Thoracic Aorta; Aneurysm Thoracic; Pseudo-aneurysm, Thoracic; Dissection of Thoracic Aorta; Intramural Haematoma of Thoracic Aorta; Penetrating Ulcer of Aorta (Disorder); Rupture of the Isthmus
Keywords: Aorta, thoracic; Aortic arch; Aorta, descending; Thoracic aortic aneurysm; Thoracic aortic dissection; Thoracic aortic stent; TAAA
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Dissection, Thoracic Aorta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Stent treatment of thoracic aortic pathologies, including aneurysms, pseudo-aneurysms, dissections, intramural hematomas, penetrating ulcers and ruptures of the isthmus, seems to provide a likely benefit compared to surgery in terms of surgical mortality and severe morbidity. However, the data concerning the long-term fate of these stents are insufficient. For this reason, the French National Health Authority (HAS) requests a 5-year follow-up in relation to the renewal of insurance reimbursement for these stent-grafts. Therefore, this long-term observational study has been set up.

DETAILED DESCRIPTION:
Study outline:

French observational, prospective, multi-center, non-randomized, single arm and open-label study.

Study device:

RELAY PLUS and RELAY NBS PLUS thoracic aortic stent or future range extension models, excluding custom-made devices.

A total of 160 patients will be included in France consecutively from all participating centers and among users of the studied stent-graft (all of the centers) or any new center during the inclusion period. The patient will be considered as included in the study when the RELAY PLUS or RELAY NBS PLUS stent-graft is introduced via the surgical or percutaneous approach and provided that the patient meets all of the study eligibility criteria.

The primary endpoint of this study is the 5-year mortality rate (all causes). The objective will be to assess the interest of the technique in terms of the long-term efficacy and safety of the use of the RELAY PLUS or RELAY NBS PLUS stent-graft (i.e. at 5 years) on a cohort of patients representative of the population treated under actual conditions of use.

The implantation of the RELAY PLUS or RELAY NBS PLUS thoracic aortic stent-graft must be carried out in accordance with recommendations issued by the Haute Autorité de Santé (HAS) including:

* Carrying out the implantation in centers with expertise in both endovascular and surgical treatments, and with an adequate technical platform.
* The implementation of a multidisciplinary discussion, in particular on the risk of surgical conversion and the possible use of cardiopulmonary bypass (CPB).
* Verification of the presence of a proximal neck of at least 2 cm in length, allowing for the stent to be placed.
* The need to educate patients about the advantages and disadvantages of the repair techniques available, such as open surgery and endo-aortic stent (EAS).
* Annual monitoring by CT-scan with contrast, or MRI + x-ray.

As this study is observational, no specific examination or procedure outside the framework of the current practice of each center is required.

A summary report will be submitted annually to the Haute Autorité de Santé (HAS). The final report was submitted on 31July2024

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring the placement of the RELAY PLUS or RELAY NBS PLUS thoracic aortic stent-graft for the treatment of a pathology of their descending thoracic aorta.
* Patient (or legal representative for minor patients) who does not object (in writing or verbally) to the collection and transmission of their data.

Exclusion Criteria:

* Patients for whom clinical follow-up is not possible, i.e. patients who are unable to return for follow-up visits (for example patients living abroad).
* Patient who earlier benefited from one or more thoracic stent-grafts and for whom a specific follow-up of the RELAY PLUS or RELAY NBS PLUS stent-graft would not be possible depending on the nature of their treatment (e.g. patient already treated with stent-graft in the descending and/or thoraco-abdominal aorta with several extensions) .

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 160 eligible patients presenting a pathology of their descending thoracic aorta and having an indication for endovascular treatment of this pathology by the RELAY PLUS or RELAY NBS PLUS thoracic aortic stent-graft will be included consecutively in this observational study. The eligibility criteria will be limited in order to best represent the population treated under real conditions of use.
  The consecutive recruitment will be carried out in all the centers using the studied stent-graft.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Long-term all-cause mortality | Any death occurring between the surgery when the stent-graft is introduced through the arterial access and the last follow-up at 5 years

SECONDARY OUTCOMES:
Rate of exclusion of the aneurysm, penetrating aortic ulcer, false channel or rupture site, with no endoleak of any type | Postoperatively or in the month following the intervention, 1 year, 2 years, 3 years, 4 years, 5 years
Rate of neurological complications | Postoperatively or in the month following the intervention, 1 year, 2 years, 3 years, 4 years, 5 years
Rate of cardiac, renal and pulmonary complications | Postoperatively or in the month following the intervention, 1 year, 2 years, 3 years, 4 years, 5 years
Rate of device-related complications | Postoperatively or in the month following the intervention, 1 year, 2 years, 3 years, 4 years, 5 years
Surgical conversion rate | Postoperatively or in the month following the intervention, 1 year, 2 years, 3 years, 4 years, 5 years
Secondary procedure rate | Postoperatively, 1 year, 2 years, 3 years, 4 years, 5 years
Pathology-related mortality rate | Postoperatively or in the month following the intervention, 1 year, 2 years, 3 years, 4 years, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pr. Pascal Desgranges, Principal Investigator — Henri Mondor Hospital, Creteil, France
Locations (10):
- France (10):
  - Hôpital Cardio-Vasculaire et Pneumologique Louis Pradel - HCL, Bron
  - CHU de Créteil - Hôpital Henri Mondor, Créteil
  - Hôpital Edouard Herriot - HCL, Lyon
  - Hôpital Européen Georges Pompidou, Paris
  - CHU de Bordeaux - Hôpital Haut Lévêque, Pessac
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne
  - Hôpitaux Universitaires de Strasbourg - NHC, Strasbourg
  - Clinique du Tonkin, Villeurbanne